CLINICAL TRIAL: NCT00088426
Title: Clinical and Genetic Studies on Holoprosencephaly
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040093; 04-HG-0093
Record Dates: First submitted 2004-07-23; First posted 2004-07-26 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Holoprosencephaly; HPE; Developmental Delay Disorders; Brain Disorders
Keywords: GENETIC DISEASE; Multiple Abnormalies; Birth Defects; Holoprosencephaly; HPE
MeSH Terms: conditions — Holoprosencephaly; Developmental Disabilities; Brain Diseases; Genetic Diseases, Inborn; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Control group of Williams-Beuren (also known as Williams) syndrome
- Family: Direct blood relatives (typically parents, and occasionally siblings of affected individuals) ofpatients with HPE are also eligible to participate.
- HPE: Patients with HPE

SUMMARY:
This study will examine how holoprosencephaly (HPE) affects people, how they change over time, and what genes may be involved in the cause of the disorder. HPE is a defect of brain development in utero in which the forebrain fails to sufficiently divide into two hemispheres, resulting in a single-lobed brain and skull and facial malformations. In most cases, the defects are so severe that babies die before birth. There are three classifications of HPE. In alobar HPE the brain does not divide at all; this form is usually associated with severe facial deformities. In semilobar HPE the hemispheres divide somewhat, causing an intermediate form of the disorder. In lobar HPE, the mildest form, separation of hemispheres is nearly normal.

Patients with HPE and their direct blood relatives may participate in this study. Patients are seen by a team of medical specialists at the NIH Clinical Center for the following procedures:

* Physical and neurological examination
* Eye examination
* Imaging studies, such as echocardiogram, abdominal ultrasound, brain MRI
* Electroencephalogram (EEG)
* Hearing evaluation
* Blood and urine samples for genetic and endocrine studies, routine blood chemistries, urinalysis, and urine electrolytes
* Other consultations as needed
* Possibly photographs, including front and side views of the face and other body parts that may be involved in HPE, such as the eyes, teeth, hands, and feet

Parents will be asked questions about the child's prenatal, birth, newborn, and past medical history, growth, behavior and development, and therapy and medication.

Because HPE is a genetic disorder and gene changes can be passed on in a family, parents will also be asked to undergo the following procedures:

* Completion of a medical and family history form
* Physical and neurological examination
* Blood and urine samples (for mothers only)
* Specialty consultations as indicated
* Possibly photographs, including front and side views of the face and other body parts that may be involved in HPE, such as the eyes, teeth, hands, and feet
* Psychosocial study. Some parents will be asked to participate in a telephone interview or complete a questionnaire, or both, about their attitudes, beliefs, and concerns about how they and their family cope with their child's condition. Some questionnaires may include questions about aspects of their marriage and personal feelings and experiences.

Parents will meet with a doctor and a genetics nurse to discuss the results of the tests and answer questions. Parents may be asked to bring their child back to the NIH after 2 years for follow-up examination and possible additional or repeat testing.

...

DETAILED DESCRIPTION:
Holoprosencephaly (HPE) is a defect of midline forebrain development that occurs soon after conception. It has a prevalence of 1 in 250 during early embryonic development, and 1 in 10,000 to 1 in 20,000 at term. In live born infants, the abnormalities associated with HPE are divided into three main categories: alobar, semilobar, and lobar HPE. A fourth variant, middle interhemispheric variant, has also been recognized. The purpose of this study is to increase our understanding of the genetic and clinical manifestations of HPE through detailed physical, psychological, developmental, neurologic, endocrinologic, and radiologic studies. We will examine the spectrum of clinical characteristics of HPE to facilitate early diagnosis and clinical management, including genetic counseling. Finally, we plan to assess the psychosocial impact of HPE on the family as a unit. Most patients and their families will be seen at the NIH Clinical Center. A subset may be examined outside the NIH, and a further subset, for the psychosocial studies, may be interviewed by phone.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Depending on their willingness to participate, subjects may enroll in DNA laboratory-only (98-HG-0249), psychosocial-only, or clinical-only. However, to conserve resources and meet study objectives, subjects with known mutations will be given priority in selection for extensive clinical studies. All races and genders are known to be at risk for HPE, anywhere in the world. Nationality or place of origin is not specific barrier to participation.
  2. Direct blood relatives (typically parents, and occasionally siblings of affected individuals) of patients with HPE are also eligible to participate.

EXCLUSION CRITERIA:

1. Anyone unwilling to provide informed consent (for themselves as adults, or on behalf of their children as minors) or assent.
2. Medical condition(s) or mental retardation are not in themselves reason for exclusion if in the judgment of the referring physician this would involve no more than minimal risk. We anticipate that children with mental handicaps would be included in the research population. We will make every effort to explain the study for the purpose of assent in a manner that the family feels is both age and developmentally appropriate for that child.
3. We generally review a brief clinical description from the referring physician about a potential research subject to determine that the subject is appropriate to enter into the study. We reserve the right to exclude cases that are clearly not HPE or related to our direct research interests (e.g. HPE cases that are syndromic like Smith Lemli Opitz syndrome, Trisomy 13, Trisomy 18, drug-related, or teratogen-related). This almost never happens, and we would attempt to make referrals to a more appropriate investigator.

It is our intention to try to remove as many economic, cultural, geographic, racial, and gender barriers as we reasonably can to promote participation of HPE cases for research purposes.

Description and justification of clinical inclusion/exclusion criteria for environmental study arm control group (individuals with Williams syndrome) :

Participants must have a confirmed diagnosis of Williams syndrome caused by deletions in chromosome 7q11 involving the Williams-Beuren Syndrome Critical Region (WBSCR). Children should be less than 6 years of age to allow for improved maternal recall of prenatal

environmental exposures. The Williams syndrome cohort (PI: Dr. Beth Kozel; National Heart Lung Blood Institute) was chosen to allow for inherent biases in mothers who have children with multiple anomaly syndromes.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with known or suspected holoprosencephaly (HPE). To conserve resources and meet study objectives, subjects with known mutations will be given priority in selection for extensive clinical studies. Direct blood relatives (typically parents, and occasionally siblings of affected individuals) of patients with HPE are also eligible to participate.@@@
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2004-01-23 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
To characterize the physical, developmental, neurologic, endocrinologic and radiologic phenotype of HPE through this comprehensive natural history study. | Once with possible followup at Year 2
  To characterize the physical, developmental, neurologic, endocrinologic and radiologic phenotype of HPE through this comprehensive natural history study.
To examine the spectrum of clinical characteristics of HPE and facilitate early clinical recognition, diagnostic confirmation, anticipatory management, prognostication, and proper genetic counseling. | Once with possible followup at Year 2
  (a) To compare gene mutations (with known or suspected abnormal functional effects) with the phenotypes observed in patients (i.e genotype-phenotype correlations) as documented in the study. (b) To determine the spectrum of brain malformations caused by genetic changes in HPE candidate genes that are known or suspected to cause human disease. (c) To correlate neurodevelopmental status/clinical outcome with neuroradiologic findings and genetic changes in HPE candidate genes. (d) To verify recurrence risks /inheritance patterns of HPE for each of the HPE candidate genes.
To determine the spectrum of non-neurologic anomalies resulting from mutations in HPE-associated genes /pathways both in individuals with HPE and individuals without HPE. | Once with possible followup at Year 2
  (a) To determine the association between mutations in HPE-associated genes/pathways and the non- neurologic finding of fatty liver in individuals with HPE. (b) To determine the presence of other, previously unknown clinical manifestations in individuals with HPE.
To assess the psychosocial impact of HPE on the family system. | Once with possible followup at Year 2
  (a) To describe characteristics of stress and coping in families of children affected by HPE. (b) To examine the relationships between specific child characteristics (e.g., chronological age, severity of disorder), family coping styles and family variables (e.g., stress, coping, marital satisfaction, parental anxiety and depression).(c) To examine the similarities and/or differences between mothers and fathers experiences of stress and coping in families of children with HPE. (d) To generate data for the development of a new instrument to quantify stress, coping and resilience in HPE families.

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Kruszka, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Golden JA. Holoprosencephaly: a defect in brain patterning. J Neuropathol Exp Neurol. 1998 Nov;57(11):991-9. doi: 10.1097/00005072-199811000-00001. No abstract available. PMID 9825935
- [Background] Matsunaga E, Shiota K. Holoprosencephaly in human embryos: epidemiologic studies of 150 cases. Teratology. 1977 Dec;16(3):261-72. doi: 10.1002/tera.1420160304. PMID 594909
- [Background] Roach E, Demyer W, Conneally PM, Palmer C, Merritt AD. Holoprosencephaly: birth data, benetic and demographic analyses of 30 families. Birth Defects Orig Artic Ser. 1975;11(2):294-313. PMID 1227533
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2004-HG-0093.html